CLINICAL TRIAL: NCT06034665
Title: Estimation of The Minimal Clinically Important Difference (MCID) for Commonly Used Outcome Measures in Patients With Knee Osteoarthritis
Brief Title: Estimation of the MCID for Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Derya Celik, Professor, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DR2022
Record Dates: First submitted 2023-05-22; First posted 2023-09-13 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; mcid; exercise; rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Other): All patients will receive an exercise rehabilitation program tailored to their needs.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — All patients will be included in the exercise program for their symptoms regarding knee osteoarthritis for 15 sessions.

SUMMARY:
Background: The effect of exercise on knee osteoarthritis (OA) is often evaluated with patient-reported scales. The Minimal Clinically Important Difference (MCID) values of these scales are needed to understand the change in patients after treatment and to manage the treatment.

It is also one of the most important data in calculating the MCID sample size. Aim: In the literature, MCID studies for exercise applied to knee OA are limited especially for those who did not undergo surgery. Thus new studies are needed.

Method: 100 patients who were diagnosed with knee osteoarthritis will be recruited for the study. Participants will be included in an exercise program tailored to their needs for 15 sessions. WOMAC, OKS, LEFS scales will be used also knee range of motion will be assessed in the baseline, after treatments and in the 4th month follow up.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with knee OA according to the criteria of the American Society of Rheumatology (ACR) (Diagnosis of primary knee OA)
* Stage 2 or 3 according to Kellgren Lawrence radiological staging criteria
* Participants with age between 50 and 70 years old
* Being able to walk without using an assistive device
* Having a body mass index of less than 30 kg/m²
* Pain severity is between 3 and 7 according to the Numerical Pain Rating Scale

Exclusion Criteria:

* Patients who received physical therapy or intra-articular injections in the last 6 months
* Receiving an indication for surgery
* Have severe hearing, vision and speech impairment
* Having serious systemic and cardiovascular diseases that interfere with exercise
* Having a lower extremity deformity
* Patients with acute inflammation of the knee

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
WOMAC | Baseline, after 15 session and 4 months follow up
  Western Ontario and McMaster Universities Osteoarthritis Index
KOOS | Baseline, after 15 session and 4 months follow up
  Knee Injury and Osteoarthritis Outcome Score
LEFS | Baseline, after 15 session and 4 months follow up
  Lower Extremity Functional Scale
Knee Range of Motion | Baseline, after 15 session and 4 months follow up
  Range of motion assessment with goniometer

SECONDARY OUTCOMES:
30s sit to stand test | Baseline, after 15 session and 4 months follow up
  For functional assessment, patient sit and stand for 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University Physiotherapy and Rehabilitation Application and Research Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No